CLINICAL TRIAL: NCT07029763
Title: Assessment of Functional Outcomes Following Successful Finger Replantation
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Talaat Ahmed, Egypt, Sohag, Elmaragha, Sohag University
Other Study IDs: Soh-Med-25-5_2MD
Record Dates: First submitted 2025-06-02; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Finger Replantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The functional outcomes following finger replantation are assessed using a combination of objective measures such as grip strength, range of motion, and sensory testing and subjective evaluations, such as patient-reported outcomes regarding pain, satisfaction, and ability to perform daily activities. Various scoring systems have been developed to standardize the assessment of these outcomes, but differences in methodology, patient demographics, and injury types often make direct comparisons difficult. Despite these challenges, it remains clear that the benefits of replantation extend beyond simply salvaging the digit; the restoration of function is a key determinant in the success of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffered traumatic digit injuries leading to total amputation as defined by Biemer (Biemer, 1980).
* Multiple digit replantation.

Exclusion Criteria:

* Multiple level amputations.
* Bad general condition.
* Mutilating hand injuries.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A prospective study will be conducted including all patients who have undergone successful finger replantation following traumatic amputations at the Plastic and Reconstructive Surgery Department, Sohag University Hospital between April 2025 and October 2026 with a follow up period at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Range of motion (ROM) | At least 6 months after replantation
  A goniometer will be used to determine the range of motion (ROM) of the metacarpophalangeal and interphalangeal joints of the replanted digits.
Finger flexion and extension of replanted digits | At least 6 months after replantation
  The fingertip-to-palm distance (FPD) and fingertip-to-table distance (FTD) will be used to assess deficits in finger flexion and extension of replanted digits.
Grip and pinch strengths | At least 6 months after replantation
  Jamar hand dynamometer will be used to determine the grip and pinch strengths. Grip and pinch measurements will be taken in the standardized sitting position with the shoulder of the patient kept in the neutral position and the elbow flexed to 90°.
Recovery of sensibility | At least 6 months after replantation
  The static two-point discrimination (2-PD) and Semmes-Weinstein monofilament test (SWM test) will be used to evaluate the sensory recovery of the radial and ulnar digital nerves of all injured fingers. Normal sensibility is defined as the sensibility assessed at the corresponding contralateral uninjured digits. The two-point discriminator consists of a plate with several pins with adjustable separations ranging from 1 to 15 mm in steps of 1 mm. The patients will be asked to close their eyes during the examination. One or two pins will be applied perpendicularly to the radial and ulnar finger pulp and held for at least 3 seconds. Three repeated responses will be necessary for the final score.
Pain intensity | At least 6 months after replantation
  Only patients with a single-digit injury will be included for these evaluations. This is because patients with multiple-digit injuries will be expected to have a higher pain level than patients with a single-digit injury and their inclusion would, therefore, bias the results. On a scale from 0 to 10, the pain intensity at rest, under strain, and in cold temperatures will be reported, with a higher number indicating increased pain.
DASH score | At least 6 months after replantation
  The disability of the arm, shoulder, and hand (DASH) questionnaire will be used for subjective evaluations. Only patients with a single-digit injury will be included for these evaluations. This is because patients with multiple-digit injuries will be expected to have a higher DASH score than patients with a single-digit injury and their inclusion would, therefore, bias the results. The DASH questionnaire contains 30 questions on daily living activities for assessing the patient's disabilities in the upper extremities. Each question is scored on a five-point scale from 1 to 5. The score calculation ranged from 0 to 100, while a higher DASH score indicated increased disability. At least 27 of the 30 items will be needed to obtain a valid score.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt